CLINICAL TRIAL: NCT06380413
Title: Effects of a 12-week Tai Chi Chuan Combined With Walking Program on Physical and Mental Parameters of Older Adults: A Randomized Controlled Trial
Brief Title: Tai Chi Chuan Combined With Walking on Physical and Mental Parameters of Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 78972024.7.0000.5313
Record Dates: First submitted 2024-04-17; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Aging
Keywords: physical exercise; tai chi chuan; walking; muscle strength; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Tai Ji; Walking

STUDY DESIGN:
Intervention Model Description: This study is a randomized, single-blinded, two-arm, parallel, superiority trial. Forty healthy and physically inactive subjects, 60 to 75 years of age, are recruited. Participants are randomly allocated on a 1:1 ratio to a 12-week intervention of Tai Chi Chuan plus walking program twice a week, or an active-control group of walking twice a week.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be implemented for the outcome assessors. All tests and questionnaires will be supervised by an evaluator blinded to the participant's group. Due to the type of intervention, the investigator conducting exercise sessions and participants will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Chuan Plus Walking (Experimental): Tai Chi Chuan plus walking program twice a week
  Interventions: Other: Tai Chi Chuan Plus Walking
- Walking (Active Comparator): Walking program twice a week
  Interventions: Other: Walking

INTERVENTIONS:
Other: Tai Chi Chuan Plus Walking — Participants perform a 12-week program with two weekly sessions on non-consecutive days. The sessions last 75 min (5 min of warm-up, 45 min of Tai Chi Chuan (TCC), 20 min of walking, and 5 min of cool-down). The intervention occurs at the School of Physical Education, Federal University of Pelotas. The TCC section occurs in a mirrored dance studio, while walking occurs on an indoor sports court. The TCC sections are based on the simplified Yang 16-movement form. Over the 12 weeks, participants learn the fundamentals and basic principles of TCC and practice the 16 movements. In the walking sections, the intensity of the effort and recovery periods are controlled through the Rate of Perceived Exertion (RPE) using the Borg scale 6-20. Effort and recovery periods are on 13 and 11 RPE, respectively. The effort and recovery lengths vary over the weeks. The training sessions are collective, with 5 to 20 participants, supervised by two experienced instructors, a TCC and a fitness instructor.
  Arms: Tai Chi Chuan Plus Walking
Other: Walking — Participants perform a 12-week training program with two weekly exercise sessions on non-consecutive days. The sessions last 30 minutes (5 minutes of warm-up, 20 minutes of walking, and 5 minutes of cool-down) throughout the intervention period. The intervention occurs in an indoor sports court at the School of Physical Education, Federal University of Pelotas. In the walking sections, the intensity of the effort and recovery periods are controlled through the Rate of Perceived Exertion (RPE) using the Borg scale 6-20. Effort and recovery periods are on 13 and 11 RPE, respectively. The effort and recovery lengths vary over the weeks. The training sessions are collective, with 5 to 20 participants, supervised by two experienced instructors, a TCC and a fitness instructor.
  Arms: Walking

SUMMARY:
Background: Tai Chi Chuan, a Chinese martial art style, is a mind-body modality that has shown positive impacts on health markers in various populations, particularly older adults. This study aims to investigate the effects of a 12-week program of Tai Chi Chuan exercises based on the Yang 16-movement form and walking on older adults' physical and mental markers.

Methods: This study is a randomized, single-blinded, two-arm, parallel, superiority trial. Forty older adults between 60 and 75 years old who are not engaged in any systematic strength and aerobic training program will be recruited. Candidates with language and cognitive problems, a history of cardiovascular diseases (except controlled hypertension), osteoarticular limitations and fractures, severe injuries, and prosthetic placement in the last six months will be excluded. Participants will be randomly allocated on a 1:1 ratio to a 12-week intervention with Tai Chi Chuan and walking two times per week, or an active-control group with walking two times per week. Physical measures will be muscle strength (i.e., knee extensors maximum strength and lower limbs functional performance -primary outcomes-, dynamic knee extensors endurance, handgrip strength, back-leg-chest strength), functional capacity, static balance, muscle thickness and muscle quality of quadriceps. Mental measures will be quality of life, sleep quality, cognitive function, and depressive and anxiety symptoms. Outcomes will be measured before and after 12 weeks of intervention. The analysis plan will use an intention-to-treat approach and protocol criteria.

Discussion: The conceptual hypothesis is that the intervention training program with Tai Chi Chuan and walking will lead to greater improvements in both physical and mental parameters due to its multi-component character compared to the walking active-control group.

ELIGIBILITY:
Inclusion Criteria:

* Not be engaged in any regular and systematic strength and aerobic training with a frequency greater than one session per week in the previous six months;
* To live in Pelotas without the intention of moving or traveling during the intervention period.

Exclusion Criteria:

* Language and cognition problems (accessed through the Mini-Mental State Examination, minimum score ≥28 points for people with >11 years of schooling, ≥23 points for people with 1-11 years of schooling, and ≥16 points for illiterate);
* History of cardiovascular diseases (except medication-controlled hypertension);
* Osteoarticular limitations that may impair physical exercise performance, such as fracture, prosthesis placement, or severe injury in the last six months.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximal dynamic strength | Baseline (week 0) to post-training (week 13)
  The maximum dynamic muscle strength of knee extensors will be measured through the one-repetition maximal test (1RM) performed in an extension chair. The 1RM value is considered the greatest load that the participant could lift for one complete repetition (i.e., concentric and eccentric phase) following a predetermined cadence (i.e., approximately 2 s per phase) controlled by a digital app (Metronome). The 1RM of each participant is determined within five attempts, and at least 3 min of rest interval was given between trials. A new load was estimated using correction factors (Lombardi, 1989) for the subsequent trial when the participant could perform more than one complete repetition. The test is rescheduled if the value of 1RM is not determined between the five attempts. According to a previous study from our laboratory (Andrade et al. 2020), the range of motion is individualized for each participant and controlled by a range of motion custom-build device.
Functional test - 30-s Chair-stand test | Baseline (week 0) to post-training (week 13)
  The 30-s Chair-Stand test is performed to measure the strength of the lower limbs. Participants are instructed to sit and stand up from a chair 43 cm high from the seat, without the aid of the upper limbs, as many times as possible during 30 s.

SECONDARY OUTCOMES:
Dynamic muscular endurance | Baseline (week 0) to post-training (week 13)
  The same knee extension machine is used to assess dynamic muscular endurance. To do so, participants perform the maximal number of bilateral knee extension repetitions at 60% of their 1RM. The test cadence (2 s for each contraction phase) and range of motion are the same for the 1RM test. The post-intervention assessment is performed using the same absolute load employed at baseline (i.e., 60% of baseline 1RM).
Isometric handgrip strength | Baseline (week 0) to post-training (week 13)
  The Handgrip isometric strength will be accessed using a handgrip dynamometer (Jamar, Sammons Preston Inc.®). Participants must be seated and with the elbow of the limb to be evaluated flexed at 90° without any external support. Both hands will be measured. On command, participants must squeeze the dynamometer as hard as possible for 5 seconds. Three attempts will be made for each hand, with a 1-minute interval between attempts, and the highest value achieved will be recorded, which is measured in Kilogram-Force (kgf).
Isometric back-leg-chest strength | Baseline (week 0) to post-training (week 13)
  The isometric back-leg-chest strength will be accessed using the back-leg-chest dynamometer (Crown, Oswaldo Filizola Ltda.), as illustrated in Figure 19. Participants must position themselves on the equipment platform with their knees extended, hips flexed at approximately 60 degrees, hands holding the equipment bar, and look straight ahead. On command, participants must pull the dynamometer upwards, exerting as much force as possible. Three attempts will be made with a 1-minute interval between attempts, and the highest value achieved will be recorded, which is measured in Kilogram-Force (kg).
Functional tests - arm curl | Baseline (week 0) to post-training (week 13)
  The Arm Curl test is performed to measure the strength of the upper limbs. Starting at full elbow extension and holding a 2 kg dumbbell in each hand, participants are instructed to perform the maximal number of elbow crunches over the full range of motion for 30 s. The test is performed with both upper limbs.
Functional tests - 8-ft Up-and-Go | Baseline (week 0) to post-training (week 13)
  The 8-ft Up-and-Go test is performed to measure agility and dynamic balance. Participants are instructed to get up from the chair (43 cm), turn around a marker that will be 2.44m, and return to the starting position. The shortest time of two attempts will be considered as a result.
Functional tests - Chair Sit-and-Reach | Baseline (week 0) to post-training (week 13)
  The Chair Sit-and-Reach test is performed to measure the flexibility of the lower limbs. Participants sit on the front edge of a chair and extend one leg straight out in front of the hip, with foot flexed and heel resting on the floor (the other leg is bent, foot flat on the floor). The object is to reach as far forward as possible toward (or past) the toes. The investigator uses a ruler noting the cm left to reach the toe (negative score) or the cm that went past the toe (positive score).
Functional tests - Back Scratch | Baseline (week 0) to post-training (week 13)
  The Back Scratch test is performed to measure the flexibility of the upper limbs. Participants are instructed to try to touch the middle fingers of both hands together behind the back. The investigator uses a ruler noting the cm left to reach the middle fingers (negative score) or the cm that the middle fingers overlapped (positive score).
Funcional tests - 6-min Walk | Baseline (week 0) to post-training (week 13)
  The 6-min Walk test is performed to measure aerobic fitness. The course proposed in the original test is 45.72 m rectangular. The course will be adapted for a straight line with 30 m length, demarcated with cones every 3 m. Participants are instructed to walk for 6-min in a flat 30m course, in which the total distance walked "as fast as possible" is assessed.
Static balance - 30-second single-leg stance test | Baseline (week 0) to post-training (week 13)
  The static balance will be determined through the 30-second single-leg stance test (Briggs et al., 1989). The subjects will be positioned facing the wall, at a distance at which they can rest their hands on the wall at shoulder height with their elbows extended. They will be asked to choose one of their lower limbs, whichever they feel most comfortable balancing on. At the signal, they will be asked to look at a fixed point on the wall, lower their upper limbs, keeping them glued to the body in an orthostatic position, and flex the knee of the lower limb not chosen to approximately 90 degrees, remaining in single-leg support. Three attempts will be made, and the longest time (30 s maximum) that participants are able to maintain a single-leg balance will be recorded.
Quadriceps muscle thickness | Baseline (week 0) to post-training (week 13)
  Transversal images of the four portions of the quadriceps femoris are obtained by B-mode ultrasonography with a 7.5 megahertz linear array probe. Images of the vastus lateralis (VL), rectus femoris (RF), and vastus intermedius (VI) muscles are obtained at the midpoint between the anterosuperior iliac spine and the upper edge of the patella, whereas the vastus medialis (VM) is assessed at 30% of the distance between the lateral condyle and the greater trochanter of the femur. All images will be analyzed using the ImageJ software (National Institutes of Health, USA, version 1.37). The muscle thickness will be assessed as the distance from each muscle's superior and inferior muscle aponeurosis. Overall quadriceps femoris muscle thickness will be calculated as the sum of each muscle thickness (i.e., RF + VL + VM + VI).
Quadriceps muscle quality | Baseline (week 0) to post-training (week 13)
  Transversal images of the four portions of the quadriceps femoris are obtained by B-mode ultrasonography with a 7.5 megahertz linear array probe. Images of the VL, RF, and VI muscles are obtained at the midpoint between the anterosuperior iliac spine and the upper edge of the patella, whereas the VM is assessed at 30% of the distance between the lateral condyle and the greater trochanter of the femur. All images will be analyzed using the ImageJ software. Muscle quality will be determined by the echo intensity values, which will be calculated from gray-scale analysis using the standard histogram function in ImageJ. The echo intensity of the quadriceps femoris will be calculated as the mean of echo intensity values of the four individual quadriceps femoris muscles ((RF + VL + VM + VI)/4).
Objective cognitive function - Trail Making Test (TMT) | Baseline (week 0) to post-training (week 13)
  Aspects of objective cognitive function are measured by the Trail Making Test (TMT). The version validated for the Brazilian population of TMT (Carvalho & Caramelli, 2020) is used to assess domains such as attention, motor skills, processing speed and cognitive flexibility (Bowie & Harvey, 2006). In the first part of the instrument (TMT-A), participants will have to draw a line connecting the numbers from 1 to 25 in ascending order. Then, letters (A-L) will be added so that the participants trace a line again following a numerical (1-13) and alphabetical order, interleaved (TMT-B). Participants will be instructed to maintain pencil-to-paper contact during the test. A shorter runtime indicates better performance.
Objective cognitive function - Controlled Oral Word Association Test (COWAT) | Baseline (week 0) to post-training (week 13)
  Aspects of objective cognitive function are also measured by the Controlled Oral Word Association Test (COWAT). The COWAT is used to assess verbal fluency, working memory and inhibitory control (Ross et al., 2007). In this test the participants will have to speak as many words as possible that start with the letters "F", "A" and "S", within 1 minute for each letter. Proper names, repeated words and variations in gender, number and conjugation will not be considered. The greater number of words evoked in each test indicates better verbal fluency.
Quality of Life - Abbreviated World Health Organization Quality of Life (WHOQOL-Bref) | Baseline (week 0) to post-training (week 13)
  Quality of life will be measured using the Abbreviated World Health Organization Quality of Life (WHOQOL-Bref) questionnaire, a validated version in Brazilian Portuguese (Fleck et al., 2000). The questionnaire has 26 questions, two general questions about quality of life, and 24 divided into four domains with six questions each: physical, psychological, social relationships, and environment.
Sleep quality - Pittsburgh Sleep Quality Index | Baseline (week 0) to post-training (week 13)
  The participants' perceived sleep quality will be measured using the Pittsburgh Sleep Quality Index, a validated version in Brazilian Portuguese (Passos et al., 2017). The questionnaire has 19 self-rated questions and five questions rated by the bed partner or roommate (if any) that investigate the quality and possible sleep disturbances during the last month across seven domains: subjective quality, sleep latency, sleep duration, sleep efficiency, sleep disorders, medication use, and daily dysfunction. Each domain has a score that varies from 0 to 3 points, totaling a maximum of 21 points. Scores above 5 points indicate poor sleep quality. The questions evaluated by the partner/colleague are not considered when calculating the final score and, for logistical reasons, will be removed from the data collection instrument.
Depressive and anxiety symptoms is measured using the Hospital Anxiety and Depression Scale (HADS) | Baseline (week 0) to post-training (week 13)
  HADS was developed by Zigmond and Snaith (1983), with translation and validation for the Brazilian population (Botega et al., 1995). It is an instrument composed of 14 items, seven of which form the anxiety subscale and the other seven the depression subscale, allowing the assessment of symptoms in the previous week. Each HADS item has four response options ranging from 0 to 3, reaching a maximum of 21 points in each subscale.

OTHER OUTCOMES:
Body mass | Baseline (week 0)
  Body mass measurements are performed using a digital scale with a stadiometer (WELMY, Santa Bárbara d'Oeste - São Paulo, Brazil). Body mass is measured in kilograms.
Height | Baseline (week 0)
  Height measurements are performed using a digital scale with a stadiometer (WELMY, Santa Bárbara d'Oeste - São Paulo, Brazil). Height is measured in meters.
Waist and hip circumferences | Baseline (week 0)
  Waist and hip circumferences are measured with a measuring tape placed around the navel height and the width of the participants' hips, respectively, to calculate the waist-hip ratio.
Monitoring the intensity of training sessions - Borg Category-Ratio 10 (CR-10) | Intervention period (week 1 to week 12)
  The intensity participants perceive in each training session will be recorded using the perceived exertion index at the end. The validated Brazilian Portuguese version of Borg's Category-Ratio 10 scale, adapted by Foster et al. (2001), will be used. The scale has values from 0 to 10, anchored to intensities of perceived effort, with 0 being equivalent to no effort (rest) and 10 to maximum effort.
Follow-up questionnaire | Post-training (week 13)
  Each participant answers 14 questions about individual perception related to the intervention using a Likert scale of 7 points, in which "1" means "no totally agreement" and "7" means "totally agreement". The questionnaire will be applied post-intervention to evaluate important outcomes in cancer patients such as safety, fun, motivation, future, benefits for daily life, intervention partner influence, training-related exhaustion, satisfaction, self-confidence on physical performance, supervision preference, changes in lifestyle, including physical activity and eating habits, and main barriers to group participation.
Adherence assessments | Intervention period (week 1 to week 12)
  (percentage of sessions attended about the total number of sessions).
Health Questionnaire | Baseline (week 0)
  A standardized questionnaire will examine aspects linked to health history, illnesses, and medication use, among other things. This questionnaire will be administered before signing the consent form to determine the eligibility of potential participants.
Level of physical activity - International Physical Activity Questionnaire (IPAQ) - extended version | Baseline (week 0)
  The extended version of the International Physical Activity Questionnaire (IPAQ) (Matsudo et al., 2001) will be used to assess the participant's level of physical activity. This questionnaire will be administered before the consent form is signed. Participants are classified as low, medium, or high according to the frequency and time of physical activity reported.
Cognitive screening - Mini-mental state examination (MMSE) | Baseline (week 0)
  The Mini-Mental State Examination will be applied to assess cognitive status (Melo; Barbosa, 2015). This questionnaire will be administered before signing the consent form to determine the eligibility of potential participants. A score of ≥28 points for people with >11 years of schooling, ≥23 points for people with 1-11 years of schooling and ≥16 points for illiterates) will be adopted as eligibility criteria (Folstein; Folstein; McHugh, 1975).

CONTACTS AND LOCATIONS:
Overall Officials: Cristine L Alberton, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Escola Superior de Educação Física e FIsioterapia, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasconcelos BB, Freitas MP, Crochemore-Silva I, Alberton CL. Effects of a 12-week Tai Chi Chuan combined with walking program on physical and mental parameters of older adults: rationale and methodological protocol for a randomized controlled trial. Trials. 2025 Oct 27;26(1):446. doi: 10.1186/s13063-025-09190-1. PMID 41146306